CLINICAL TRIAL: NCT03622450
Title: The Effect of Colistin Inhalation on the Clinical Outcome of Patients With Ventilator Associated Pneumonia
Brief Title: The Effect of Colistin Inhalation on Ventilator Associated Pneumonia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nourhan Hassan Osama Thuraya Mohamed (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Nourhan Hassan Osama Thuraya Mohamed, Clinical pharmacist, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Colistin inhalation form
Record Dates: First submitted 2018-06-18; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Colistin; Carbapenems; Aminoglycosides; Quinolones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medication arm (Experimental): Colistin to be given as 2 millions three times daily in the inhalation form from 5 to 7 days in addition to another antipseudomonal antibiotic according to infectious disease society of antimicrobials (IDSA) guidelines from day 1 of incidence of ventilator associated pneumonia
  Interventions: Drug: Colistin
- Control arm (Active Comparator): Patients receive antipseudomonal antibiotics IV as carbapenem and quinolone or aminoglycoside according to IDSA guidelines from day 1 of incidence of Ventilator associated pneumonia carbapenem as 1g three times daily + tavanic 750mg once daily or ciprofloxacin 500mg twice daily or aminoglycoside according to renal function
  Interventions: Drug: Carbapenem + Aminoglycoside/ Quinolone

INTERVENTIONS:
Drug: Colistin — Polymyxins are bactericidal drugs that bind to lipopolysaccharides (LPS) and phospholipids in the outer cell membrane of gram-negative bacteria.
  Other Names: Colomycin
  Arms: Medication arm
Drug: Carbapenem + Aminoglycoside/ Quinolone — Dual antipseudomonal given as IV for ventilator associated pneumonia for patients with Multi-drug resistant bacteria risk factors
  Other Names: tienam,meropenem,levofloxacin,ciprofloxacin,amikacin,gentamicin
  Arms: Control arm

SUMMARY:
The study has been conducted to measure the clinical outcome of early intervention with colistin inhalation in patients with ventilator associated pneumonia suspected to have multidrug resistant gram -ve bacteria

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years

Patients presenting with signs of infection 48 hours of intubation

Exclusion Criteria:

* Patients with documented bronchiectasis

Cystic fibrosis Known allergy to polymyxin. Patients presenting with chest infection or signs of infection before intubation.

Patients with creatinine clearance less than 30ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2018-01-06 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Assessment of Ventilatory status | 7 to 10 days
  Pf ratio measurement

SECONDARY OUTCOMES:
Days of mechanical ventilation | 35 Days
  Deescalation in the ventilation mode and trials until successful weaning.
Time till the occurence of sepsis | 35 Days
  long standing ventilator associated pneumonia with failure of treatment can lead to sepsis
Mortality as an outcome of long stand untreatable ventilator associated pneumonia | 35 days
  is the mortality due to sepsis of other causes
Length of stay in the icu | 35 days
  How long will the patient stay in the ICU according to failure of weaning and progression of the disease.

IPD SHARING:
Plan to Share IPD: No
Number of patients ,statistical data, method,discussion and outcome will be shared